CLINICAL TRIAL: NCT05433441
Title: Evaluation of the Effectiveness of the Parkinson's Specialized Teams Intervention on the Quality of Life of Parkinson's Patients in the Territory of the Nouvelle-Aquitaine and Hauts-de-France: ES-Park Pilot Study.
Brief Title: Evaluation of the Effectiveness of the Parkinson Specialized Teams Intervention
Acronym: ES-Park
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CHUBX 2022/02
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease
Keywords: Parkinson; Quality of life; Complementary non drug intervention; Multidisciplinary approach
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (No Intervention)
- ESPark Intervention (Experimental): Under medical prescription and in addition to medical and physiotherapy care, the ESPark will intervene in an ecological way with Parkinson's patients in order to rehabilitate them, maintain their autonomy in their daily life and their social life with the aim of improving the quality of life of the patient and his main caregiver. Beyond a rehabilitative intervention in the home, the ESPark's mission would also be to optimize the patient's living environment and possibly help with the implementation of the necessary aids in the continuity of medical care.
  Interventions: Procedure: ESPark Intervention

INTERVENTIONS:
Procedure: ESPark Intervention — The treatment will include 15 sessions (1 session per week). An initial assessment will be carried out during the first session in order to determine the objectives and the personalized follow-up.
  Arms: ESPark Intervention

SUMMARY:
A pilot experiment interventional study is proposed in order to set up multidisciplinary team for Parkinson's patients at home. The aim of this study is to evaluate the effectiveness of this specialized Parkinson's team (ESPark) intervention a on the quality of life of patients with moderate to severe Parkinson's disease

DETAILED DESCRIPTION:
Parkinson's disease (PD) and related disorders are the second most common cause of motor disability in the elderly after stroke. Progressively, the disability impacts the activities of daily living and social life of Parkinson's patients with a major impact on their quality of life. The diversity and complexity of the needs of parkinsonian patients and their caregivers justify a specific multidisciplinary approach. Several studies have evaluated the effectiveness of the intervention of such teams on the maintenance of activities of daily living and quality of life of Parkinson's patients with contradictory results. In France, the experience of specialized Alzheimer teams (ESA) based on the same concept seems to have brought positive results on autonomy and resocialization. Based on the positive experience of ESA intervention in Alzheimer's disease and in view of the data in the literature on Parkinson's disease, we would like to develop the same type of care with teams adapted to the problems of Parkinson's disease patients, which we could call ESParks, and to evaluate the effectiveness of such teams in the context of support for Parkinson's patients.

ELIGIBILITY:
Inclusion Criteria:

For the patient:

* Patient with a diagnosis of idiopathic Parkinson's disease
* Patient over 18 years ;
* Patient with a Hoehn and Yahr Stage greater than or equal to 3;
* Patient without major cognitive impairment defined by a MOCA score ≥21
* Patient living at home ;
* Patient with an identified non-professional primary caregiver;
* Person affiliated with or benefiting from a social security plan;
* Free, informed and and express consent (confirmed in writing) (no later than the day of inclusion and before any examination required by the research).

For the caregiver:

* Male or female over 18 years
* Able to respond to research interviews/questionnaires
* Free, informed and express consent (confirmed in writing) (no later than the day of inclusion and before any examination required by the research).

Exclusion Criteria:

For the patient:

* Patient with medically indicated dementia impairing comprehension and adherence, and/or with severe confusion or psycho-hallucinatory state;
* Institutionalized or foster care patients;
* Patients with a known severe and unstable general pathology that does not allow for patient follow-up;
* Patients already included in another non-drug management trial;
* Patients whose institutionalization is envisaged in the short term (within 6 months) or for whom a change of residence is envisaged in the short term and would not allow for follow-up assessments;
* Patients under guardianship or unable to express consent
* Primary caregiver not wishing to participate in the study or unable to be available for the planned study follow-up;
* Presence of a primary caregiver with a known severe and unstable disease that does not allow for the conduct of the study;
* Presence of a primary caregiver with a known cognitive or psychiatric disorder (chronic progressive psychosis) that does not allow for the proper conduct of the study.
* Pregnant or breastfeeding woman.

For the caregiver:

* Unable to follow the research interviews or questionnaires.
* Primary caregiver not wishing to participate in the study or unable to be available for the planned study follow-up;
* Primary caregiver with a known severe and unstable illness that does not allow for the proper conduct of the study;
* Primary caregiver with known cognitive or psychiatric disorders (chronic progressive psychosis) that do not allow the study to be conducted properly.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-12-06 (Actual); Primary Completion 2025-12-06 (Estimated); Study Completion 2027-06-06 (Estimated)

PRIMARY OUTCOMES:
Score of quality of life scale (PDQ 39) | Initial Visit - Day 0
  Self-questionnaire in 39 items evaluating the quality of life of Parkinson's patients from a motor and psychological point of view. Each question is rated from 0 (no disturbance) to 4 (maximum disturbance). The items are divided into 8 dimensions (activity of daily living, emotional well-being, psychological discomfort, social support, cognitive impairment, communication, physical discomfort, mobility) It consists of 39 items with a total score that varies from 0 to 154
Score of quality of life scale (PDQ 39) | 6 months
  Self-questionnaire in 39 items evaluating the quality of life of Parkinson's patients from a motor and psychological point of view. Each question is rated from 0 (no disturbance) to 4 (maximum disturbance). The items are divided into 8 dimensions (activity of daily living, emotional well-being, psychological discomfort, social support, cognitive impairment, communication, physical discomfort, mobility) It consists of 39 items with a total score that varies from 0 to 154

SECONDARY OUTCOMES:
IADL assessment | Initial Visit - Day 0
  Assessment of the level of dependence in instrumental activities of daily living It consists of 9 items with a total score that varies from 0 to 36 Each item is scored from 0 (autonom) to 4 (no autonom) or NA
IADL assessment | 6 months
  Assessment of the level of dependence in instrumental activities of daily living
IADL assessment | 12 months
  Assessment of the level of dependence in instrumental activities of daily living
Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Rate | Initial Visit - Day 0
  Used to evaluate the various motor and non-motor symptoms. In this protocol, only motor examination will be carried out. This part includes the following items: speech, facial expression, rigidity, finger tapping, hand movements, hand pronation supination movements, toe tapping, leg agility, getting up from the examination chair, walking, postural stability, posture, overall spontaneity of movement, postural hand tremor, hand action tremor, amplitude of resting tremor, constancy of resting tremor. The items of the Parkinsonian triad are evaluated on the different parts of the body (extremities of the limbs, lip and jaw for resting tremor and neck for rigidity). The presence of dyskinesias is mentioned at the end of the evaluation and if they interfered with the motor examination, as well as the global scale of Hoehn and Yahr. All items are rated from 0 to 4 and are clearly defined : 0: normal, 1 = minimal, 2 = mild, 3 = moderate, 4 = severe
Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Rate | 6 months
  Used to evaluate the various motor and non-motor symptoms. In this protocol, only motor examination will be carried out. This part includes the following items: speech, facial expression, rigidity, finger tapping, hand movements, hand pronation supination movements, toe tapping, leg agility, getting up from the examination chair, walking, postural stability, posture, overall spontaneity of movement, postural hand tremor, hand action tremor, amplitude of resting tremor, constancy of resting tremor. The items of the Parkinsonian triad are evaluated on the different parts of the body (extremities of the limbs, lip and jaw for resting tremor and neck for rigidity). The presence of dyskinesias is mentioned at the end of the evaluation and if they interfered with the motor examination, as well as the global scale of Hoehn and Yahr. All items are rated from 0 to 4 and are clearly defined : 0: normal, 1 = minimal, 2 = mild, 3 = moderate, 4 = severe
Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Rate | 12 months
  Used to evaluate the various motor and non-motor symptoms. In this protocol, only motor examination will be carried out. This part includes the following items: speech, facial expression, rigidity, finger tapping, hand movements, hand pronation supination movements, toe tapping, leg agility, getting up from the examination chair, walking, postural stability, posture, overall spontaneity of movement, postural hand tremor, hand action tremor, amplitude of resting tremor, constancy of resting tremor. The items of the Parkinsonian triad are evaluated on the different parts of the body (extremities of the limbs, lip and jaw for resting tremor and neck for rigidity). The presence of dyskinesias is mentioned at the end of the evaluation and if they interfered with the motor examination, as well as the global scale of Hoehn and Yahr. All items are rated from 0 to 4 and are clearly defined : 0: normal, 1 = minimal, 2 = mild, 3 = moderate, 4 = severe
Non-motor symptoms Scale for Parkinson's Disease (NMSS) | Initial Visit - Day 0
  30-item scale that assesses a wide range of non-motor symptoms in patients with Parkinson's disease (PD). The NMSS measures the severity and frequency of non-motor symptoms across nine dimensions. The scale can be used for patients in all stages of PD.
Non-motor symptoms Scale for Parkinson's Disease (NMSS) | 6 months
  30-item scale that assesses a wide range of non-motor symptoms in patients with Parkinson's disease (PD). The NMSS measures the severity and frequency of non-motor symptoms across nine dimensions. The scale can be used for patients in all stages of PD.
Non-motor symptoms Scale for Parkinson's Disease (NMSS) score | 12 months
  30-item scale that assesses a wide range of non-motor symptoms in patients with Parkinson's disease (PD). The NMSS measures the severity and frequency of non-motor symptoms across nine dimensions. The scale can be used for patients in all stages of PD.
Montreal Cognitive Assessment (MOCA) score | Initial Visit - Day 0
  The MoCA assesses mild cognitive dysfunction. It assesses the following functions: short-term memory, visual-spatial skills, executive functions, attention, concentration, working memory, language, abstraction, calculation and orientation in time and space. Cognitive impairment is assessed using a 30-point score (27-30: no cognitive impairment; 18-26: mild; 10-17: moderate; < 10: severe).
Montreal Cognitive Assessment (MOCA) score | 6 months
  The MoCA assesses mild cognitive dysfunction. It assesses the following functions: short-term memory, visual-spatial skills, executive functions, attention, concentration, working memory, language, abstraction, calculation and orientation in time and space. Cognitive impairment is assessed using a 30-point score (27-30: no cognitive impairment; 18-26: mild; 10-17: moderate; < 10: severe).
Montreal Cognitive Assessment (MOCA) score | 12 months
  The MoCA assesses mild cognitive dysfunction. It assesses the following functions: short-term memory, visual-spatial skills, executive functions, attention, concentration, working memory, language, abstraction, calculation and orientation in time and space. Cognitive impairment is assessed using a 30-point score (27-30: no cognitive impairment; 18-26: mild; 10-17: moderate; < 10: severe).
Beck Depression Inventory (BDI-II) score | Initial Visit - Day 0
  Self-questionnaire comprising a list of 21 items measuring the somatic, affective and cognitive severity of depressive symptoms. Each item is rated for symptom severity and/or frequency, over the past 7 days, on a 4-point scale ranging from 0 to 3. Higher scores indicate severe symptomatology.
Beck Depression Inventory (BDI-II) score | 6 months
  Self-questionnaire comprising a list of 21 items measuring the somatic, affective and cognitive severity of depressive symptoms. Each item is rated for symptom severity and/or frequency, over the past 7 days, on a 4-point scale ranging from 0 to 3. Higher scores indicate severe symptomatology.
Beck Depression Inventory (BDI-II) score | 12 months
  Self-questionnaire comprising a list of 21 items measuring the somatic, affective and cognitive severity of depressive symptoms. Each item is rated for symptom severity and/or frequency, over the past 7 days, on a 4-point scale ranging from 0 to 3. Higher scores indicate severe symptomatology.
Parkinson Anxiety Scale (PAS) Score | Initial Visit - Day 0
  Self-questionnaire assessing anxiety in Parkinson's disease dealing with several dimensions of anxiety: Persistent anxiety (5 items), Episodic anxiety (4 items), Avoidance behavior (3 items). Each item is scored from 0 (not at all) to 4 (strongly or almost always).
Parkinson Anxiety Scale (PAS) Score | 6 months
  Self-questionnaire assessing anxiety in Parkinson's disease dealing with several dimensions of anxiety: Persistent anxiety (5 items), Episodic anxiety (4 items), Avoidance behavior (3 items). Each item is scored from 0 (not at all) to 4 (strongly or almost always).
Parkinson Anxiety Scale (PAS) Score | 12 months
  Self-questionnaire assessing anxiety in Parkinson's disease dealing with several dimensions of anxiety: Persistent anxiety (5 items), Episodic anxiety (4 items), Avoidance behavior (3 items). Each item is scored from 0 (not at all) to 4 (strongly or almost always).
Reduced Neuropsychiatric Inventory (NPI-R) score | Initial Visit - Day 0
  Used to assesses 12 domains of psychobehavioral disorders (21). It is a questionnaire consisting of a screening question and seven to nine items for each of the 12 domains: delusions, hallucinations, agitation/aggressiveness, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, motor aberration, behavioural disorders, sleep, appetite and eating. The score ranges from 0 to 144 .
Reduced Neuropsychiatric Inventory (NPI-R) score | 6 months
  Used to assesses 12 domains of psychobehavioral disorders (21). It is a questionnaire consisting of a screening question and seven to nine items for each of the 12 domains: delusions, hallucinations, agitation/aggressiveness, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, motor aberration, behavioural disorders, sleep, appetite and eating. The score ranges from 0 to 144 .
Reduced Neuropsychiatric Inventory (NPI-R) score | 12 months
  Used to assesses 12 domains of psychobehavioral disorders. It is a questionnaire consisting of a screening question and seven to nine items for each of the 12 domains: delusions, hallucinations, agitation/aggressiveness, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, motor aberration, behavioural disorders, sleep, appetite and eating. The score ranges from 0 to 144 .
Zarit scale score | Initial Visit - Day 0
  This scale assesses caregiver burden ; it consists of 22 items with a total score that varies from 0 to 88. (score ≤20, no burden - score> 60, severe burden).
Zarit scale score | 6 Months
  This scale assesses caregiver burden ; it consists of 22 items with a total score that varies from 0 to 88. (score ≤20, no burden - score> 60, severe burden).
Zarit scale score | 12 Months
  This scale assesses caregiver burden ; it consists of 22 items with a total score that varies from 0 to 88. (score ≤20, no burden - score> 60, severe burden).
State Trait Anxiety Inventory short scale (STAI-E and STAI-T) score | Initial Visit - Day 0
  This anxiety scale consists of 2 scales of 20 questions that assess how subjects feel at the time and generally.
State Trait Anxiety Inventory short scale (STAI-E and STAI-T) score | 6 months
  This anxiety scale consists of 2 scales of 20 questions that assess how subjects feel at the time and generally.
State Trait Anxiety Inventory short scale (STAI-E and STAI-T) score | 12 months
  This anxiety scale consists of 2 scales of 20 questions that assess how subjects feel at the time and generally.
Quality of life as measured by the PQoL Carers. | Initial Visit - Day 0
  Quality of life questionnaire for caregivers Self-questionnaire comprising a list of 26 items with a total score that varies from 0 to 104
Quality of life as measured by the PQoL Carers. | 6 months
  Quality of life questionnaire for caregivers Self-questionnaire comprising a list of 26 items with a total score that varies from 0 to 104
Quality of life as measured by the PQoL Carers. | 12 months
  Quality of life questionnaire for caregivers Self-questionnaire comprising a list of 26 items with a total score that varies from 0 to 104
Sense of competence questionnaire | Initial Visit - Day 0
  This 35-item questionnaire covers three areas: the impact of caregiving on the caregiver's personal life, satisfaction with one's own performance as a caregiver, and satisfaction with the person with dementia as a recipient of care Each item is scored from 1 ("yes") to 3 ("No") and 2 (Yes/no) The total score varies from 27 to 81
Sense of competence questionnaire | 6 months
  This 35-item questionnaire covers three areas: the impact of caregiving on the caregiver's personal life, satisfaction with one's own performance as a caregiver, and satisfaction with the person with dementia as a recipient of care Each item is scored from 1 ("yes") to 3 ("No") and 2 (Yes/no) The total score varies from 27 to 81
Sense of competence questionnaire | 12 months
  This 35-item questionnaire covers three areas: the impact of caregiving on the caregiver's personal life, satisfaction with one's own performance as a caregiver, and satisfaction with the person with dementia as a recipient of care Each item is scored from 1 ("yes") to 3 ("No") and 2 (Yes/no) The total score varies from 27 to 81
Ressource Utilization in Dementia (RUD) | Initial Visit - Day 0
  The questionnaire allows us to estimate the medico-social costs associated with the care of the patient. This estimate is based on the evaluation of the quantity of formal resources (including social services, home care) and informal resources (care and assistance provided by the caregiver) involved in the day-to-day care of the patient; the resources are valued economically using the health insurance rates, where applicable, and the hourly costs of medical and social assistance at home
Ressource Utilization in Dementia (RUD) | 6 Months
  The questionnaire allows us to estimate the medico-social costs associated with the care of the patient. This estimate is based on the evaluation of the quantity of formal resources (including social services, home care) and informal resources (care and assistance provided by the caregiver) involved in the day-to-day care of the patient; the resources are valued economically using the health insurance rates, where applicable, and the hourly costs of medical and social assistance at home
Ressource Utilization in Dementia (RUD) | 12 Months
  The questionnaire allows us to estimate the medico-social costs associated with the care of the patient. This estimate is based on the evaluation of the quantity of formal resources (including social services, home care) and informal resources (care and assistance provided by the caregiver) involved in the day-to-day care of the patient; the resources are valued economically using the health insurance rates, where applicable, and the hourly costs of medical and social assistance at home

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra FOUBERT-SAMIER, Principal Investigator — University Hospital, Bordeaux
Locations (4):
- France (4):
  - Hopital Pellegrin, Bordeaux
  - CHU de Lille, Lille
  - CHU de Limoges, Limoges
  - CHU Poitiers, Poitiers